CLINICAL TRIAL: NCT03706248
Title: Evaluation of the Performance and Sensitivity of the Clinical Genomics Colvera Test in Predicting Recurrence of Colorectal Cancer
Brief Title: Paired Analysis of Sensitivity for Colorectal Cancer Using COLVERA : PASCAL
Acronym: PASCAL
Status: Completed | Type: Observational
Sponsor: Clinical Genomics Pathology (Industry)
Responsible Party: Sponsor
Other Study IDs: CG0013
Record Dates: First submitted 2018-10-11; First posted 2018-10-15 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If there is leftover plasma, the plasma or the DNA extracted from the plasma may be stored at the sponsor for repeat assays.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No recurrence: CT scan has confirmed that subjects are without recurrence. Blood can be drawn up to 4 weeks after scan.
  Effective Feb 28, 2019, this group is closed to accrual as it has reached the goal.
  Interventions: Other: Blood Draw
- Recurrence: CT scan has confirmed that subjects are have recurrence of their colorectal cancer. Blood can be drawn prior to any treatment for the recurrent disease.
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw — 20 ml of blood will be drawn from subjects via venipuncture

SUMMARY:
To compare the sensitivity and specificity estimates of Colvera with that of a commercially available CEA test for detection of recurrent disease in subjects with colorectal cancer that have documented recurrence or no evidence of recurrence by CT.

DETAILED DESCRIPTION:
The study will be carried out as a single cohort, observational, prospective study to compare sensitivity of Colvera to detect recurrent colorectal cancer confirmed by radiology imaging (CT) with CEA sensitivity in paired testing. Blood is collected for assay of methylated BCAT1 and IKZF1 DNA and CEA, from subjects who have undergone curative treatment for primary CRC of stages II and III (AJCC) and who are in remission (No evidence of disease). Subjects will have recently (within 4 weeks of blood collection) had follow-up radiological imaging as part of their surveillance program for recurrence. Participation is for one visit only as part of each subject's surveillance-monitoring schedule. Two PAXgene blood tubes (minimum 10 mL, maximum 20 mL) will be collected. Any evidence of methylated BCAT1 and/or IKZF1 DNA in blood represents a Colvera "positive" result. CEA levels of 5ug/L or higher will represent a "positive" result. Sensitivity and specificity of the Colvera and CEA test will be estimated and compared in a paired fashion in each case where recurrence status has been investigated and determined by the site clinical management team. Blood testing shall be performed and analyzed by qualified staff blinded to clinical status. This is a cross-sectional observational non-significant risk study, and test results will not be used for clinical management, i.e. there will be no interventions in subjects consenting to participate in this Research Study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older, and capable and willing to provide informed consent.
2. Subject has undergone curative treatment for primary CRC of stages II and III (AJCC).
3. Subject was determined to be in remission at the conclusion of primary therapy and has been in clinical surveillance for at least 6 months. (No imaging is required for the determination of remission. Last treatment was at least 6 months earlier. No requirement to complete all of the initial adjuvant treatment plan.)
4. Subject has had a surveillance CT scan within the past 4 weeks and either has recurrent CRC or does not have recurrent CRC based on that CT scan result.
5. Subject is willing to provide a blood sample. (2 PAXgene tubes)
6. Definition of recurrence is evidence of local tumor recurrence or metastasis by CT scan of chest, abdomen and pelvis or other modalities that confirm recurrent CRC

Exclusion Criteria:

1. Subject has other cancer at the time of recruitment.
2. Subject has prior history of recurrent CRC.
3. Subject has a diagnosis of End Stage Renal Disease (ESRD), with or without current dialysis treatment.
4. Subject's life expectancy is less than one year based on performance status and clinical signs and symptoms.
5. Subject is receiving chemo- or radiotherapy at the time of blood collection, or between radiological imaging and blood collection.
6. Results of the recent surveillance CT of the chest, abdomen and pelvis are inconclusive regarding recurrence of CRC, and further work up (other imaging and/or biopsy) is not required at this time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective study will enroll 50 subjects with radiologic confirmation of recurrence of colorectal cancer and 50 subjects without CRC recurrence (documented by CT scan). Eligible study subjects will include men and women (18 years or older) of any race and ethnicity who have completed treatment (no further adjuvant chemotherapy or surgery currently planned) for primary CRC of stages II and III (AJCC, [2]), and have been considered by the site clinical management team for at least 6 months to be in remission. . (Concurrent imaging is not required as part of the clinical determination of remission. Subjects who have had a recent (within 4 weeks) or prior CT scan for purposes of surveillance are eligible.)
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2018-07-28 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive predictive value and negative predictive value | 1 year
  Comparison of Colvera and CEA in recurrent and non-recurrent CRC

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Torrance Memorial Physician Network, Redondo Beach, California
  - University of South Florida, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Colon and Rectal Surgery Associates, Metairie, Louisiana
  - Providence Hospital-Ascension Health, Novi, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Data from each subject is captured without any identifiers in an electronic database.
Supporting Information: Study Protocol, SAP, ICF, CSR